CLINICAL TRIAL: NCT00004206
Title: Phase II Study of Oxaliplatin and 5 Fluorouracil in the Treatment of Advanced Ovarian Cancer
Brief Title: Oxaliplatin and Fluorouracil in Treating Patients With Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067452; LRI-IND.02-V3; EU-99036
Record Dates: First submitted 2000-01-21; First posted 2003-11-04 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining oxaliplatin and fluorouracil in treating patients who have recurrent ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of oxaliplatin in combination with fluorouracil in terms of response rate, time to tumor progression, and overall survival in patients with recurrent ovarian cancer. II. Evaluate the safety profile of this combination regimen in this patient population.

OUTLINE: This is an open label study. Patients receive oxaliplatin IV over 2 hours once every 2 weeks and fluorouracil IV and leucovorin calcium IV once weekly. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease are followed at 1 month and at 3 months, then every 3 months for disease relapse and survival.

PROJECTED ACCRUAL: A total of 14-50 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ovarian cancer Must have received at least one prior platinum based chemotherapy regimen and have relapsed within 2 years of last chemotherapy regimen Evaluable disease Radiology confirmation AND/OR Elevated CA 125 (at least 60 IU/L)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) (unless documented Gilbert's syndrome) AST/ALT less than 3 times ULN (less than 5 times ULN if liver metastases present) Renal: Creatinine normal Cardiovascular: No unstable cardiovascular disease Other: No active, uncontrolled infection No other significant medical disorder or condition that would preclude study No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified Other: At least 30 days since prior investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth O'Byrne, MD, Study Chair — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, England, United Kingdom